CLINICAL TRIAL: NCT02217176
Title: Ultrasonography of the Neck: The Influence of Airway Devices on Vascular Topography in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Harran University (Other)
Responsible Party: Principal Investigator, Menekse Ozcelik, Specialist of Anesthesiology and Intensive Care Medicine, Ankara University
Other Study IDs: 31-662
Record Dates: First submitted 2014-08-10; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Ultrasonography, Pediatrics, Overlap, Vascular Structures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- endotracheal intubation
- laryngeal mask airway

SUMMARY:
Internal jugular venous catheterization is a challenging procedure in pediatric patients due to small size. Overlapping of the internal jugular vein (IJV) and common carotid artery (CCA) may jeopardize the success and increase the complication rate.However, the use of ultrasound as an assistance tool might be helpful to identify the relationship between the IJV and the CCA. Endotracheal intubation and insertion of laryngeal mask are the common options for the airway management during general anesthesia for central venous catheterization. In this observational study, the investigators aimed to investigate the impact of the laryngeal mask insertion or endotracheal intubation and the role of head rotation on the overlap of the IJV and CCA evaluated with ultrasound in pediatric patients undergoing any kind of surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologist status I-IV

Exclusion Criteria:

* patients with prior internal jugular vein catheterization or cardiovascular system anomaly

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The pediatric population who were undergone any type of surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the overlap percentages (%) of right and left IJVs before and just after insertion of LMA compared with ETT. Overlap percentage is calculated as overlap of IJV(mm)/carotid artery diameter(mm))*100 obtained from ultrasonographic images. | Obtaining ultrasonographic images takes 30 minutes on average per patient
  The airway devices are identified according to the own preference of the responsible anesthesiologist regarding to the patient's status and the type of surgery.
  Ultrasonographic images of each patient are recorded bilaterally with a 8-12 MHz linear probe (Venue 40 GE, USA) at the cricoid cartilage level perpendicular to the skin, parallel to mandibula in neutral, 40o and 80o head away position. The same ultrasonographic evaluations are repeated after the airway device insertion. The images are then evaluated by three different anesthesiologist.

SECONDARY OUTCOMES:
the relationship between IJV and CCA defined as anterior, anterolateral, lateral, anteromedial and medial according to the IJV's topographic location | Obtaining ultrasonographic images takes 30 minutes on average per patient

OTHER OUTCOMES:
the diameter of bilateral IJVs in mm | Obtaining ultrasonographic images takes 30 minutes on average per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Department of Anesthesiology and Intensive Care Medicine, Ankara, Turkey (Türkiye)